CLINICAL TRIAL: NCT06537999
Title: A Phase 2, Randomized, Double-Blinded, Placebo-Controlled, Study to Evaluate Safety, Tolerability, Pharmacometrics, and Efficacy of DNTH103 in Adults With Multifocal Motor Neuropathy (MOMENTUM)
Brief Title: A Clinical Study to Evaluate DNTH103 in Adults With Multifocal Motor Neuropathy
Acronym: MOMENTUM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dianthus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNTH103-MMN-201; 2024-513128-40-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Multifocal Motor Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DNTH103 low dose Q2W (Experimental)
  Interventions: Drug: DNTH103
- DNTH103 high dose Q2W (Experimental)
  Interventions: Drug: DNTH103

INTERVENTIONS:
Drug: DNTH103 — * Day 1: IV loading dose
  * Week 1 to Week 15: DNTH103 administered SC every 2 weeks
  Other Names: Claseprubart
  Arms: DNTH103 high dose Q2W; DNTH103 low dose Q2W
Drug: Placebo — * Day 1: IV infusion of placebo
  * Week 1 to Week 15: placebo administered SC every 2 weeks
  Arms: Placebo

SUMMARY:
The purpose of this Phase 2 study is to evaluate the safety, tolerability, pharmacometrics, and efficacy of DNTH103 in participants with multifocal motor neuropathy (MMN).

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out
2. Adult males and females, 18 to 75 years of age (inclusive).
3. Weight range between 40 to 120 kilograms (kg).
4. Confirmed diagnosis of definite or probable MMN.
5. Evidence of:

   1. Responsiveness to Ig treatment; and
   2. Receiving a stable Ig regimen
6. Documented vaccinations against encapsulated bacteria in accordance with local requirements and vaccine availability.
7. Female participants must be of nonchildbearing potential or if of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use a highly effective method of contraception.
8. Male participants must be surgically sterile for at least 90 days prior to Screening or agree not to donate sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable method of contraception.

Exclusion Criteria:

1. History or presence of significant medical/surgical condition including any acute illness or major surgery considered to be clinically significant or that could impact efficacy assessments.
2. Any coexisting conditions which may interfere with outcome assessments (eg, severe diabetic neuropathy).
3. Concurrent or previous use of rituximab, cyclophosphamide, mycophenolate mofetil, azathioprine, or cyclosporine. If a participant has previously used these medications, the last dose must be at least 6 months prior to randomization.
4. Currently or previously on complement inhibitors including in a clinical trial setting.
5. Prior history (at any time) of N. meningitidis infection.
6. Diagnosis of an autoimmune disorder other than MMN.
7. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies during Screening.
8. History of active malignancy within 5 years prior to Screening, except basal cell carcinoma of the skin, curatively resected squamous cell carcinoma of the skin, cervical carcinoma in situ curatively treated or low-grade prostate adenocarcinoma for which appropriate management is observation alone.
9. Participation in another clinical study of an investigational drug within 90 days or 5 half-lives of the investigational agent (whichever is longer) prior to randomization (Day 1).
10. Any other overlapping condition for which the condition or treatment of the condition may affect the study assessments or outcomes.
11. Any other condition, including mental illness or prior therapy, that in the opinion of the Investigator would make the participant unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs) | Baseline to Week 17
  Incidence of treatment-emergent adverse events (TEAEs) and treatment emergent serious adverse events (SAEs)

SECONDARY OUTCOMES:
Time to Retreatment With Immunoglobulin (Ig) Since the Final Ig Treatment Before Randomization | Baseline to Week 17
  Time between the participant's last dose of Ig and when they require the next dose of Ig after entering the randomized, controlled treatment period of the study
Time to Clinical Deterioration (CD) | Baseline to Week 17
  The time it takes a participant to meet defined criteria for worsening of symptoms in the study
Mean Value, Mean Change, and Percentage Change From Baseline in Grip Strength | Baseline to Week 17
  Grip strength measured in kilopascal (kPa) using a vigorimeter
Area Under Curve (AUC) of the Change From Baseline in Grip Strength | Baseline to Week 17
  Grip strength measured in kPa using a vigorimeter
AUC of the Change From Baseline in Medical Research Council (MRC)-10 Sum Score | Baseline to Week 17
  MRC-10 evaluates motor strength/weakness from a predetermined set of 10 muscle pairs (upper and lower limbs) on a scale of 0 to 5
Mean Value and Mean Change From Baseline in MRC-10 Sum Score | Baseline to Week 17
  MRC-10 evaluates motor strength/weakness from a predetermined set of 10 muscle pairs (upper and lower limbs) on a scale of 0 to 5
Mean Value and Mean Change From Baseline in MRC-14 Sum Score | Baseline to Week 17
  MRC-14 evaluates motor strength/weakness from a predetermined set of 14 muscle pairs (upper and lower limbs) on a scale of 0 to 5
Mean Value and Mean Change From Baseline in Multifocal Motor Neuropathy Rasch-Built Overall Disability Scale (MMN-RODS) Score | Baseline to Week 17
  MMN-RODS consists of 25 items scored on a 3-point scale
Mean Value and Mean Change From Baseline in Average Time to Complete the 9-Hole Peg Test (9-HPT) | Baseline to Week 17
  9-HPT is a quantitative measure of upper extremity (arm and hand) function and dexterity
Mean Change From Baseline in Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Score | Baseline to Week 17
  INCAT comprises 2 parts, the arm score and the leg score. Each part is scored between 0 and 5 points, resulting in an INCAT total score between 0 and 10. Adjusted INCAT disability score excludes changes in upper limb function from 0 (normal) to 1 (minor symptoms)
Mean Change From Baseline in Euro-Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) Scale | Baseline to Week 17
  EQ-5D-5L is comprised of 5 dimensions: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression
Mean Change From Baseline in EQ-5D-5L Visual Analog Scale (VAS) | Baseline to Week 17
  A vertical VAS is included in the EQ 5D 5L. Participants mark their health status from 0 to 100
Count and Proportion of Participants With Patient Global Impression of Change (PGIC) Score of Improved or Better | Baseline to Week 17
  PGIC is a 7-point scale depicting a participant's rating of overall improvement
Mean Change From Baseline in Fatigue Severity Scale (FSS) Score | Baseline to Week 17
  FSS assesses disabling fatigue in participants with chronic illness
Mean Change From Baseline in Health-Related Productivity Questionnaire (HRPQ) Outcomes | Baseline to Week 17
  HRPQ is a participant diary tool designed to provide data on health-related impacts to labor force participation
Effectiveness, Side Effects, Convenience, and Overall Satisfaction Scores as Assessed by Treatment Satisfaction Questionnaire for Medications (TSQM)-14 | Baseline to Week 17
  TSQM-14 is a 14-item treatment satisfaction questionnaire that evaluates the following domains: effectiveness, side effects, convenience, and global satisfaction
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs) | Up to Week 52 of OLE
  Incidence of treatment-emergent adverse events (TEAEs) and treatment emergent serious adverse events (SAEs)
Serum Concentrations of DNTH103 | Baseline to Week 17
  Blood samples will be collected for measurement of serum concentrations of DNTH103 at various timepoints both pre- and post-dose
Incidence and Titer of Antidrug Antibody (ADA) Levels Against DNTH103 | Baseline to Week 17
  Blood samples will be collected to measure ADA against DNTH103 at various timepoints

CONTACTS AND LOCATIONS:
Locations (25):
- United States (10):
  - Clinical Study Site, Scottsdale, Arizona
  - Clinical Study Site, Los Angeles, California
  - Clinical Study Site, Bradenton, Florida
  - Clinical Study Site, Tampa, Florida
  - Clinical Study Site, Honolulu, Hawaii
  - Clinical Study Site, Kansas City, Kansas
  - Clinical Study Site, Chapel Hill, North Carolina
  - Clinical Study Site, Cincinnati, Ohio
  - Clinical Study Site, Columbus, Ohio
  - Clinical Study Site, Houston, Texas
- Denmark (2):
  - Clinical Study Site, Aarhus
  - Clinical Study Site, Copenhagen
- France (2):
  - Clinical Study Site, Marseille
  - Clinical Study Site, Paris
- Clinical Study Site, Rome, Italy
- Netherlands (2):
  - Clinical Study Site, Amsterdam
  - Clinical Study Site, Utrecht
- Clinical Study Site, Skopje, North Macedonia
- Poland (3):
  - Clinical Study Site, Bydgoszcz
  - Clinical Study Site, Katowice
  - Clinical Study Site, Krakow
- Clinical Study Site, Belgrade, Serbia
- Clinical Study Site, Barcelona, Spain
- United Kingdom (2):
  - Clinical Study Site, London, England
  - Clinical Study Site, Oxford, England